CLINICAL TRIAL: NCT04589832
Title: Phase 1B/2 Study of PAC-1 and Entrectinib for Patients With Metastatic Uveal Melanoma
Brief Title: Study of PAC-1 and Entrectinib for Patients With Metastatic Uveal Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study required dose reductions to the lower dose level (Dose level -1). But this dose level (Dose level -1) was not further explored because of lack of funding.
Sponsor: Arkadiusz Z. Dudek, MD (Other)
Collaborators: HealthPartners Institute Regions Cancer Care Center (Other); Vanquish Oncology, Inc. (Industry); Genentech, Inc. (Industry); Midwest Melanoma Partnership (Other)
Responsible Party: Sponsor-Investigator, Arkadiusz Z. Dudek, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL18-372
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Uveal Melanoma
Keywords: uveal melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — entrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Treatment Arm (Experimental): Phase 1b will determine the MTD of PAC-1 in combination with entrectinib. Study treatment will include: PAC-1 will be taken orally on Days 1-21 and Entrectinib will be taken orally on Days 1-28 of each 28-day cycle. Treatment will continue until disease progression (based on RECIST 1.1 criteria), unacceptable toxicity, subject withdrawal of informed consent, or subject death either from progression of disease, the therapy itself, or from other causes.
  Interventions: Drug: PAC-1; Drug: Entrectinib

INTERVENTIONS:
Drug: PAC-1 — Pharmacokinetic (PK) and pharmacodynamic (PD) assay for PAC-1 will be performed during Days 1 and 21 of Cycle 1. PAC-1 will be given on Day 1 of Cycle 1, withheld on Day 2 and Day 3 of Cycle 1 then reinitiated on Day 4 of Cycle 1 to continue for 21 days of the 28-day cycle. For each successive cycle, PAC-1 therapy will be initiated on Day 1 and continue for 21 days of the 28-day cycle.
Drug: Entrectinib — Pharmacokinetic and pharmacodynamic assay for entrectinib will be performed during Days 3 and 21 of Cycle 1. Entrectinib therapy will be withheld on Day 1 and Day 2 of Cycle 1, initiated on Day 3 of Cycle 1 and continue for the remainder of the 28 day cycle. For each successive cycle, entrectinib will be intiated on Day 1 and continue for 28 days of the 28-day cycle.

SUMMARY:
Single arm study with dose escalation Phase Ib cohort followed by a Phase II cohort. PAC-1 (PO) will be given daily on Days 1 through 21 of each cycle (28-day cycle). Entrectinib (PO) will be given daily on Days 1 through 28 of each cycle. Response will be evaluated after every 2 cycles. Treatment will continue until disease progression based on RECIST criteria or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately. Patients must be willing and able to provide written informed consent for this trial.
2. Age ≥ 18 years at the time of consent.
3. Histologically or cytologically confirmed metastatic uveal melanoma. Staging per AJCC manual edition 8.
4. One or more lesions that could be accurately measured using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 (Appendix 1).
6. Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 14 days prior to registration.

   * Leukocytes ≥ 2,000 µ/l
   * Absolute Neutrophil Count (ANC) ≥ 1,500 K/mm3
   * Platelets ≥ 100,000/µl
   * Hemoglobin (Hgb) ≥ 9 g/dL
   * Serum Creatinine ≤ 1.5 x ULN
   * Calculated creatinine clearance ≥ 40 mL/min
   * Total Bilirubin ≤ 1.5 mg/dL
   * Aspartate aminotransferase (AST) ≤ 2.5 × ULN
   * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
   * Alkaline Phosphatase ≤ 2.5 × ULN
   * Partial Thromboplastin Time (PTT) < 1.5 × ULN
7. Subjects must have archival tissue (metastatic disease preferred) available or undergo a biopsy prior to Cycle 1 Day 1 of treatment. Subjects that do not have archival tissue or cannot undergo a biopsy are not eligible for the study.
8. Prior therapy is allowed but must have been completed 21 days prior to initiation of protocol therapy and all toxicities must be < Grade 2.
9. Palliative radiation must have been completed 2 weeks prior to the initiation of study therapy.
10. Patient with known brain metastases must have been treated at least 2 weeks prior to enrollment, be asymptomatic from brain metastases, stable on brain imaging, and not be receiving a supra-physiologic dose of steroids (>10 mg prednisone daily or equivalent).
11. Women must not be pregnant or breastfeeding. All women of childbearing potential (WOCBP) must have a blood human chorionic gonadotrophin (hCG) test or urine hCG test within 2 weeks prior to registration to rule out pregnancy.
12. Women of childbearing potential (WOCBP) must agree to use contraception as outlined in the protocol from the time of informed consent, during the study and for 3 months after the last dose of study drug(s). Abstinence from heterosexual intercourse is an acceptable form of contraception. Women of childbearing potential are those who have not been surgically sterilized or have not been free of menses >1 year
13. Male patients who are sexually active with WOCBP must agree to use contraception as outlined in the protocol from the time of initiation of study treatment, during the study and for 3 months after the last dose of study drug(s). Abstinence from heterosexual intercourse is an acceptable form of contraception.
14. The participant is capable of understanding and complying with the protocol and has signed informed consent document.

Exclusion Criteria

1. Peripheral sensory neuropathy Grade ≥ 2 (per CTCAE v5.0).
2. Active gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would reasonably impact drug absorption.
3. Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
4. Has known active Hepatitis B or C. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay. For patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg), the patient is only eligible if they are negative for HBV DNA.
5. Known interstitial lung disease, interstitial fibrosis, or history of tyrosine kinase inhibitor-induced pneumonitis. NOTE: Radiation-induced lung disorders are not included in this exclusion criterion.
6. History of retinal pigmented epithelial detachment, central serous retinopathy, or retinal vein occlusion in the unaffected eye; or intraocular pressure 21 mmHg or uncontrolled glaucoma (irrespective of intraocular pressure) in the unaffected eye.
7. History of uncontrolled seizures.
8. History of ataxia.
9. Allergies and adverse drug reaction: History of allergy to study drug components.
10. Thromboembolic events requiring therapeutic anticoagulation. Concomitant anticoagulation with oral anticoagulants (warfarin, direct thrombin or factor Xa inhibitors), platelet inhibitors (e.g. Clopidogrel, high dose aspirin) is prohibited. Low-dose aspirin (<100 mg/day), low-dose warfarin (<1 mg/day) and prophylactic low molecular weight heparin (LMWH) or similar agent are permitted.
11. History of recent (within the past 3 months) symptomatic congestive heart failure or ejection fraction ≤ 50% observed during screening for the study.
12. History of prolonged QTc interval (e.g., repeated demonstration of a QTc interval > 450 milliseconds from ECGs performed at least 24 hours apart).
13. History of additional risk factors for torsades de pointes (e.g., family history of long QT syndrome).
14. Cardiovascular disorders including unstable angina pectoris, clinically-significant cardiac arrhythmias, myocardial infarction or stroke (including transient ischemic attack [TIA], or other ischemic event) within 6 months prior to registration.
15. Active infection requiring intravenous systemic treatment.
16. Serious non-healing wound/ulcer/bone fracture within 28 days prior to registration.
17. Known uncontrolled, symptomatic brain metastasis or cranial epidural disease.
18. Known additional malignancies which require systemic treatment.
19. Inability to swallow intact tablets.
20. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study or could compromise protocol objectives in the opinion of the Investigator and/or the sponsor-investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, PhD, Principal Investigator — Health Partners Institute
Locations (1):
- HealthPartners Institute Regions Cancer Care Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boudreau MW, Tonogai EJ, Schane CP, Xi MX, Fischer JH, Vijayakumar J, Ji Y, Tarasow TM, Fan TM, Hergenrother PJ, Dudek AZ. The combination of PAC-1 and entrectinib for the treatment of metastatic uveal melanoma. Melanoma Res. 2023 Dec 1;33(6):514-524. doi: 10.1097/CMR.0000000000000927. Epub 2023 Sep 22. PMID 37738028

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Treatment Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 63.5 [34 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Determine Maximum Tolerated Dose (MTD)
Description: The MTD of PAC-1 in combination with entrectinib is the highest tested dose of PAC-1 combined with entrectinib with DLT rate of less than 33% in first cycle of therapy (i.e., ≤1 out of 6 subjects with DLT)
Time Frame: 28 days
Population: Because of episodes of neutropenia in two patients and grade 2 dizziness and ataxia in two patients after the first cycle of therapy, dose interruptions and reductions to a lower dose level (Dose level -1: 625 mg PAC-1 + 400 mg Entrectinib) were required. The new dose level (Dose level -1) was not further explored due to lack of funding. Therefore, the study did not determine an MTD.
Measure: Number; unit: mg
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 6
mg
  PAC-1(Dose level 1) | 625
  Entrectinib(Dose level 1) | 600

2. Primary Outcome: Phase 2: Progression Free Survival at 3 Months
Description: PFS is defined as proportion of alive subjects with metastatic uveal melanoma at 3 months from treatment initiation with PAC-1 in combination with entrectinib without evidence of radiological disease progression by RECIST 1.1.
Time Frame: Time of treatment start until the criteria for disease progression.
Population: This study is terminated at phase 1b without reaching MTD due to lack of funding. Therefore, there is no accrual in phase 2.
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Assess Adverse Events
Description: The frequency and severity of all treatment related grade 1 and 2 adverse events are reported by CTCAEv5 term and grade.
Time Frame: AEs will be recorded from time of signed informed consent until 90 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 10 months.
Population: This study is terminated at phase 1b due to lack of funding. Therefore, no accrual in phase 2.
Measure: Number; unit: Participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 6
Participants
  Dizziness | 4
  Dysarthria | 4
  Anemia | 4
  Increased creatinine | 4
  Fatigue | 3
  Ataxia | 2
  Dysgeusia | 2
  Neutropenia | 2
  AST elevation | 2
  Face edema | 2
  Constipation | 2
  Skin pain | 2
  ALT elevation | 1
  Flashing lights | 1
  Eye Floaters | 1
  Tinnitus | 1
  Akathisia | 1
  Dyspepsia | 1
  Nausea | 1
  Abdominal pain | 1
  Urinary incontinence | 1
  Urinary hesitancy | 1
  Euphoria | 1
  Memory impairment | 1
  Numbness | 1
  Back pain | 1
  Edema limbs | 1
  Sensory neuropathy | 1
  Macular rash | 1
  Thrombocytopenia | 1
  Presyncope | 1
  Mental fog | 1

4. Secondary Outcome: Phase 2: Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR is defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1.
Time Frame: Start of treatment until disease progression/recurrence
Population: This study is terminated at phase 1b without reaching MTD due to lack of funding. Therefore, no accrual in phase 2 and no result available for ORR.
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 2: Duration of Response (DoR)
Description: DoR is defined as the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented
Time Frame: Time from complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease.
Population: This study is terminated at phase 1b due to lack of funding. Therefore, no accrual in phase 2 and no result for DoR.
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from treatment initiation with PAC-1 in combination with entrectinib until death as a result of any cause
Time Frame: up to a maximum of 15 months
Population: This study is terminated at phase 1b due to lack of funding. Therefore, no accrual in phase 2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 6
Months
  Phase 1b: OS | 11.49 [8.1 to 14.75]
  Phase 2: OS: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 15 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to a maximum of 10 months.
Arm/Group | Study Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment Arm (N=6)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment Arm (N=6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
AKATHISIA (Nervous system disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 4 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (5)
ATAXIA (Nervous system disorders) | 2 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHOLESTEROL HIGH (Investigations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 3 (4)
CREATININE INCREASED (Investigations) | 4 (5)
DEPRESSION (Psychiatric disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (3)
DIZZINESS (Nervous system disorders) | 4 (13)
DYSARTHRIA (Nervous system disorders) | 5 (6)
DYSGEUSIA (Nervous system disorders) | 3 (8)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
EDEMA FACE (General disorders) | 2 (2)
EDEMA LIMBS (General disorders) | 2 (3)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
EUPHORIA (Psychiatric disorders) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FATIGUE (General disorders) | 4 (4)
FEVER (General disorders) | 1 (1)
FLASHING LIGHTS (Eye disorders) | 1 (1)
FLOATERS (Eye disorders) | 1 (3)
GAIT DISTURBANCE (General disorders) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPOTENSION (Vascular disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (5)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 2 (3)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (5)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 2 (6)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (2)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (4)
WEIGHT GAIN (Investigations) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT04589832/Prot_SAP_000.pdf